CLINICAL TRIAL: NCT04301609
Title: Randomized, Comparative, Double-blind, and Placebo-controlled Clinical Trial to Assess the Improvement of Fatigue, Sleep, Anxiety / Depression, Neurovegetatives Alterations and Quality of Life After the Administration of ImmunoVita® in Chronic Fatigue Syndrome Patients
Brief Title: Clinical Trial to Assess the Improvement of Fatigue, Sleep Problems, Anxiety / Depression, Neurovegetatives Alterations and Quality of Life After the Administration of ImmunoVita® in Chronic Fatigue Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitae Health Innovation (Industry)
Collaborators: Hospital Vall d'Hebron (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PR(AG)447/2019
Record Dates: First submitted 2020-03-04; First posted 2020-03-10 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Chronic Fatigue Syndrome; Myalgic Encephalomyelitis
Keywords: Fatigue Syndrome; Encephalomyelitis; Fibromyalgia
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Encephalomyelitis; Fibromyalgia | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ImmunoVita® (Active Comparator): 250 mg Yeast beta-glucan + 3.75 microg Vitamin D3 + 1.05 mg Vitamin B6 + 7.5 mg zinc)
  Interventions: Dietary Supplement: Active
- Placebo (Placebo Comparator): 473,2 mg microcristalline cellulose + 0,06 mg Brown Oxide dye + 0,27 mg yellow A oxide dye
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Active — Take 4 capsules daily (2 capsules on an empty stomach + 2 capsules 30 minutes before dinner).
  Other Names: ImmunoVita®
  Arms: ImmunoVita®
Dietary Supplement: Placebo — Take 4 capsules daily (2 capsules on an empty stomach + 2 capsules 30 minutes before dinner).
  Arms: Placebo

SUMMARY:
Chronic Fatigue Syndrome, also known as Myalgic Encephalomyelitis (CFS / MS) is a medical entity characterized mainly by debilitating and prolonged fatigue lasting more than 6 months, post-exertion fatigue (physical and / or mental), non-sleep restorative, cognitive impairment and orthostatic intolerance with prolonged recovery that is not relieved by rest. Currently, the etiopathogenic mechanisms of the disease are not known, although mitochondrial dysfunction with bioenergetic immuno-metabolism alterations, oxidative stress, and immuno-inflammatory response stands out. At present, there is no diagnostic test, nor effective treatment in the disease. ImmunoVita, is a food supplement composed of the latest yeast beta-glucans, in addition to vitamin D3, vitamin B6 and zinc, which could contribute to the normal functioning of the immune system and the inflammatory response.

DETAILED DESCRIPTION:
In patients with CFS / ME, neuroimmune, gastrointestinal, autonomic and cardiovascular alterations have been observed, among others. CFS / ME is characterized by disabling chronic fatigue, non-restorative sleep, severe intolerance to physical exercise, neurocognitive dysfunction with changes in concentration and immediate memory and neurovegetative symptoms in the form of dizziness, syncopes and alterations in bowel and bladder rhythm . Within the etiopathogenic hypotheses of the disease, they are involved if patients treated with ImmunoVita® could significantly reduce the scores on the scale of the impact of fatigue, sleep problems, neurovegetative dysfunction, anxiety / depression, and improve the quality of life compared to the placebo group.

Based on the different etiopathogenic hypotheses of the syndrome, various mechanisms would be involved, which could modulate them, the ImmunoVita food complex.

1. Do patients with CFS / ME have high scores on the fatigue impact scale, hospital anxiety-depression scale and Pittsburg sleep quality questionnaire?
2. Do patients with CFS / ME have high scores in the autonomic dysfunction symptomatology scale?
3. Do patients with CFS / ME have low scores in the SF-36 quality of life questionnaire?
4. Do CFS / MS patients treated with ImmunoVita significantly reduce the scores on the scales of fatigue, anxiety / depression and autonomic dysfunction?
5. Will patients with CFS / ME treated with ImmunoVita significantly increase the scores on the SF-36 quality of life questionnaire?

GOALS

Main goal

The objective of this study is to assess the efficacy of active ImmunoVita® in patients with CFS / MS vs. placebo in the perception of fatigue, evaluated through the scale of perception of fatigue (FIS-40).

Secondary goals:

1. Evaluate the efficacy of active ImmunoVita® in patients with CFS / MS vs. placebo in the improvement of sleep dysfunction, through the Pittsburg questionnaire.
2. Analyze the efficacy of active ImmunoVita®, in patients with CFS / ME vs. placebo in the improvement of anxiety-depressive symptomatology, through the hospital anxiety-depression scale (HAD).
3. Evaluate the efficacy of active ImmunoVita®, in patients with CFS / ME vs. placebo in the improvement of the quality of life, through the SF-36 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both sexes, between 18-65 years.
* Patients with a BMI ≤ 25.
* Patients diagnosed with Chronic Fatigue Syndrome according to diagnostic criteria of 1994 CDC / Fukuda and 2003 Canadian criteria from the University of Central Sensitization Syndrome (Vall d'Hebron University Hospital, Barcelona).
* Patients who freely grant written consent.

Exclusion Criteria:

* Patients who are participating in another clinical trial of the same or different nature in the last 30 days prior to inclusion.
* Any subject that, in the opinion of the investigator, is not able to follow the instructions or make a good completion of the treatment.
* Subjects who do not grant written informed consent to participate in the study.
* Patients who are receiving any of the prohibited drugs or products and that the withdrawal of the drugs / products not allowed in the study is expected to pose a relevant problem.
* Pregnant women and / or during breastfeeding periods.
* Patients under treatment with oral anticoagulants.
* Patient with any type of immunosuppression.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Perception of fatigue (FIS-40). | 9 months
  The Fatigue Impact Scale (FIS-40) is a 40-item questionnaire designed to assess fatigue symptoms as part of an underlying chronic condition. It includes three domains reflecting the perceived feeling of fatigue: physical (10 items), cognitive (10 items) and psychosocial functions (20 items). Each item is scored from 0 (no fatigue) to 4 (severe fatigue). The overall score is calculated by adding together the responses to the 40 questions (ranging from 0 to 160). Higher scores indicate more functional limitations due to fatigue.

SECONDARY OUTCOMES:
Sleep dysfunction (Pittsburg questionnaire) | 9 months
  The Pittsburgh Sleep Quality Index (PSQI) is a 19-item self-administrated questionnaire commonly used to assess sleep disturbances over a 1-month interval. Scores are acquired on each of seven domains of sleep quality: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each domain is scored from 0 to 3 (0 = no problems and 3 = severe problems). The overall PSQI score ranges from 0 to 21 points, with scores of > 5 indicating poorer sleep quality.
Hospital anxiety-depression scale (HAD) | 9 months
  To assess anxiety and depression symptoms the Hospital Anxiety and Depression Scale (HADS) was used; a validated 14 item self-reported measure (seven items associated with anxiety symptoms and seven with depression) over the last week. Each item is scored on a 4-point Likert scale (e.g., 0 = as much as I always do; 1 = not quite so much; 2 = definitely not so much; and 3 = not at all) giving maximum subscale scores of 21 for depression and anxiety, respectively. Scores of 0-7 are interpreted as normal; scores of 8-10 reflect mild symptoms, 11-14 moderate, and 15-21 severe for either anxiety or depression. The global HADS score ranges from 0 (no anxiety/depression) to 42 (severe anxiety/depression).
Quality of life (SF-36) | 9 months
  The SF-36 questionnaire was used to assess health-related quality of life. This is a 36-item broadly-based self-report survey of physical and mental functioning status related to health. The SF-36 assesses functioning on eight subscales including domains of physical functioning, physical role functioning, bodily pain, general health perception, vitality, social role functioning, emotional role functioning, and mental health. Lower scores indicate a more negative impact of an individual's health on functioning.

CONTACTS AND LOCATIONS:
Overall Officials: José Alegre, PhD, Principal Investigator — Hospital Vall d´Hebron
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castro-Marrero J, Saez-Francas N, Santillo D, Alegre J. Treatment and management of chronic fatigue syndrome/myalgic encephalomyelitis: all roads lead to Rome. Br J Pharmacol. 2017 Mar;174(5):345-369. doi: 10.1111/bph.13702. Epub 2017 Feb 1. PMID 28052319
- [Background] Barbado Hernandez FJ, Gomez Cerezo J, Lopez Rodriguez M, Vazquez Rodriguez JJ. [The chronic fatigue syndrome and its diagnosis in internal medicine]. An Med Interna. 2006 May;23(5):238-44. doi: 10.4321/s0212-71992006000500009. No abstract available. Spanish. PMID 16817704
- [Background] Akramiene D, Kondrotas A, Didziapetriene J, Kevelaitis E. Effects of beta-glucans on the immune system. Medicina (Kaunas). 2007;43(8):597-606. PMID 17895634
- [Background] El Khoury D, Cuda C, Luhovyy BL, Anderson GH. Beta glucan: health benefits in obesity and metabolic syndrome. J Nutr Metab. 2012;2012:851362. doi: 10.1155/2012/851362. Epub 2011 Dec 11. PMID 22187640
- [Background] Ganda Mall JP, Casado-Bedmar M, Winberg ME, Brummer RJ, Schoultz I, Keita AV. A beta-Glucan-Based Dietary Fiber Reduces Mast Cell-Induced Hyperpermeability in Ileum From Patients With Crohn's Disease and Control Subjects. Inflamm Bowel Dis. 2017 Dec 19;24(1):166-178. doi: 10.1093/ibd/izx002. PMID 29272475